CLINICAL TRIAL: NCT01016717
Title: Clopidogrel Proton-Pump Inhibitors Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Since the published data resolved the study goals we decided not to start it
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-09-7345-MS-CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
Keywords: clopidogrel; platelet function; omeprazole; pantoprazole; coronary disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Omeprazole; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator): Patients will be taking omeprazole tablets 40 mg QD for 30 days
  Interventions: Drug: Omeprazole
- Pantoprazole (Active Comparator): Patients will be taking Pantoprazole tablets 40 mg QD for 30 days
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Omeprazole — All patients will be taking omeprazole (Losec, Abic Inc., Israel) tablets 40 mg QD for 30 days
  Other Names: Losec
  Arms: Omeprazole
Drug: Pantoprazole — Pantoprazole tablets (Controloc 40, 40 mg/day, Nycomed, Perrigo Inc., Israel). All patients will take pantoprazole tablets 40 mg QD for 30 days
  Other Names: Controloc
  Arms: Pantoprazole

SUMMARY:
To find out the impact of two different proton-pump inhibitors (PPIs) (Omeprazole and Pantoprazole) on platelet function in patients with stable coronary artery disease (CAD) on clopidogrel therapy.

DETAILED DESCRIPTION:
On June 19, 2009 The European Medicines Agency (EMEA) has issued a public statement on a possible interaction between clopidogrel (Plavix, Sanofi-Aventis/Bristol-Myers Squibb)and proton-pump inhibitors (PPIs) and has recommended that the product information for all clopidogrel-containing medicines be amended to discourage concomitant use of PPIs unless absolutely necessary. The UK medicines regulator, the Medicines and Healthcare Products Regulatory Agency (MHRA), has also issued advice to GPs that concomitant use of a PPI with clopidogrel is not recommended unless considered essential, urging a review of the prescribing of PPIs at the next appointment for patients taking clopidogrel. This follows an "early communication" issued by the US FDA earlier this year, stating that PPIs might interfere with the effectiveness of clopidogrel and that clinicians should reevaluate starting or continuing treatment with a PPI in patients taking clopidogrel.

There is a concern that the studies on which these warnings are based have many limitations and that it is far from certain whether there really is an interaction between clopidogrel and PPIs.

Another point of uncertainty is whether there may be a difference between individual PPIs, with some pharmacodynamic studies suggesting an interaction with omeprazole but not with pantoprazole. The clinical evidence, however, is conflicting. There has been one clinical trial from Canada suggesting an interaction with omeprazole but not with pantoprazole. From a mechanistic view it is known that omeprazole is metabolized by the CYP219 enzyme, which converts clopidogrel into its active metabolite. And while pantoprazole can also be metabolized by this enzyme, it also uses other routes.

Thus, the primary goal of the current study is to find out the impact of two different PPIs (Omeprazole, Losec, and Pantoprazole) on platelet function in patients with stable coronary artery disease (CAD) on clopidogrel therapy.

Forty patients with stable CAD will be randomized to receive either omeprazole tables (Losec, 40 mg/day, Abic Inc., Israel) or pantoprazole tables (Controloc 40, 40 mg/day, Nycomed, Perrigo Inc., Israel) for 1 month (Phase 1), followed by a 4-week washout period, and the alternative treatment for 1 month (Phase 2).Platelet function tests will be assessed 4 times: before and after each study phase. Following an overnight fast, ECG and blood tests for measurements of platelet function, lipids, blood cell count, electrolytes, fasting glucose, and high-sensitivity C-reactive protein (hs-CRP), will be performed. The blood samples, except those for platelet function, will be centrifuged immediately for 15 minutes at 3000/min. The sera will be stored at -20° C, and will be tested at the end of the study. Blood samples for platelet function will be assessed immediately after the blood is drawn. All blood samples will be evaluated in the same laboratory and by the same operator who will be blinded to the patients' clinical status and PPIs allocation.

All patients will be instructed to continue taking their regular medications throughout the study period. In addition, patients will be instructed not to add any medications (including over the counter medications) and to record any change in concomitant medications throughout the study period.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years; signed informed consent
2. Outpatient CAD patients on aspirin tablets 100-325 mg daily and clopidogrel tablets 75 mg daily.
3. Left ventricular (LV) systolic dysfunction ≥ 40% measured within the past 6 months.
4. No changes in cardiac medications during 2 weeks prior to enrollment.

Exclusion criteria:

1. Presence of transplanted tissue or organ or LVAD
2. AICD or CRT or CRTD patients.
3. Acute MI, CABG, PCI within past 3 months.
4. Congestive heart failure (CHF) ≥ NYHA 2.
5. Ejection fraction < 40% measured within the past 6 months.
6. Malignancy.
7. Active myocarditis, or cardiomyopathy.
8. HIV infection or immunodeficiency state.
9. Chronic viral infection.
10. Acute systemic infection requiring antibiotics.
11. Chronic diarrhea or malabsorption.
12. Statin therapy initiation ≤ 3 months.
13. Diabetes mellitus type 1.
14. Diabetes mellitus type 2 with HbA1C > 7%
15. Low-density lipoprotein cholesterol (LDL-C) > 100 mg/dL.
16. Not on statin therapy.
17. Liver function tests (LFT) ≥ x 3 upper limit of normal (ULN) or creatinine kinase (CPK) ≥ x 10 ULN.
18. Hypo/hyper thyroidism.
19. Liver dysfunction.
20. Renal failure with serum creatinine ≥ 2 mg/dL.
21. Alcohol or drug abuse.
22. Refuse to sign informed consent.
23. On the following therapy: Amiodarone, coumadin, any antibiotics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Platelet function tests. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, MA, Principal Investigator — Leviev Heart Center, Sheba Medical Center, Tel Hashomer
Locations (1):
- Leviev Heart Center, Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No